CLINICAL TRIAL: NCT05264935
Title: Ultrasound-guided Lavage of Calcific Deposits of the Rotator Cuff: The Role of Power Doppler Sonography
Brief Title: Ultrasound-guided Lavage of Calcific Deposits of the Rotator Cuff
Acronym: Kalklavage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: OE-0164
Record Dates: First submitted 2022-02-08; First posted 2022-03-03 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Rotator Cuff Tendinitis; Ultrasonography, Interventional; Ultrasonography, Doppler, Color
Keywords: calcific deposit; ultrasound-guided puncture and lavage; power doppler ultrasound
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Therapeutic Irrigation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-Guided Puncture and Lavage (UGPL) — After local anaesthesia with rapidocain the calcific deposit of the rotator cuff will be punctured and washed out with saline solution.

SUMMARY:
The primary goal of the study is to assess ultrasonographic Power Doppler signals after ultrasound-guided puncture and lavage of rotator cuff calcific tendinitis of the shoulder. Secondary outcomes are sonographic features like the course of residual calcific material and the course of tendon healing als well as the clinical symptoms of the patient.

DETAILED DESCRIPTION:
In our study we investigate the intensity of the power doppler signal after ultrasound-guided puncture and lavage (UGPL) of the rotator cuff calcific tendinitis. We assume that UGPL will lead to intratendinous neovascularisation and that the amount of retrieved calcific material is associated with the PDUS signal. The measurement of the signal will be performed in pre determined time slot for 12 months. Additional we study the correlation between the PDUS signal and the clinical symptoms of the patient and the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and older
* Pain in the deltoid region worsening with activities above shoulder level and/or at night with a calcific deposit
* Ultrasound evaluation of the calcific deposit with type I or II characteristics, a solitary conformation, a minimum size of 1.0 x 0.5 x 0.4cm (length x width x depth) and without clear signs of resorption (PDUS grade 0 - I°, see study procedure).
* In case of multiple calcific deposits, it has to be warranted that the other deposits are smaller than the minimum size of 1.0 x 0.5 x 0.4cm and with no signs of PDUS signals.
* Qualification for more intensive treatment on account of no clinical improvement after a minimum of 3 months with conservative treatment (physical therapy and oral anti-inflammatory drugs).
* able to understand the content of the patient information / consent form in German and give consent to take part in the project

Exclusion Criteria:

* Previous UGPL or surgery of the affected shoulder
* Treatment with subacromial injection (SAI) or ESWT in the three months before inclusion
* Other causes of shoulder complaints (e.g. rotator cuff tear, frozen shoulder, inflammatory arthritis, bursitis, …)
* Intervention failure (no retrieval of calcific material, leakage of the injected saline, disruption of the calcific rim or distribution of calcific material)
* Patients with a language barrier hindering questionnaire completion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with calcific deposit within the rotator cuff of a minimum size of 1.0 x 0.5 x 0.4cm (length x width x depth) and without clear signs of resorption.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
PDUS signal intensity | One year after intervention
  Power doppler ultrasonography (PDUS) signal intensity

SECONDARY OUTCOMES:
Residual calcific material | One year after intervention
  Residual calcific material (constant, decreasing, increasing)
Tendon rupture | One year after intervention
  Follow up sonography will be performed to assess the occurrence of tendon rupture, which will be classified as complete, transmural or non transmural
Pain level | One year after intervention
  Pain Scale Numeric Rating Scale from 0 (no pain) to 15 (worse pain) as part of the Constant Score
Constant Murley Score (CMS) | One year after intervention
  Constant Murley Score (CMS) from 0 (worse) to 100 (better) points
Shoulder function parameters | One year after intervention
  Shoulder range of motion (ROM) parameters in degree including elevation (flexion), abduction, and external rotation by 0° abduction measured with a standard goniometter
Shoulder function parameters | One year after intervention
  Shoulder strength in 90° abduction position (measured also for the opposite shoulder)(Kg) measured with a spring balance.
Subjective shoulder value (SSV) | One year after intervention
  Subjective shoulder value (SSV) is a patient-reported subjective outcome assessing on a scale from 0% (worse) to 100% (best) of normal shoulder condition
Level of improvement | One year after intervention
  Patients are reporting separately if the improvement / shoulder status regarding pain, function and quality of life is acceptable (Yes/No) or not for them.

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No